CLINICAL TRIAL: NCT01246167
Title: An International, Prospective, Randomized, Multicenter, Controlled Head-to-Head Comparison of Conservative, Plate Fixation and Prosthesis in Treatment of Displaced 2, 3, and 4 Part Fractures of Proximal Humerus of 60 Years and Older Patients
Brief Title: Treatment of Proximal Humeral Fractures
Acronym: TPHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Kuopio University Hospital (Other); Jyväskylä Central Hospital (Other); Karolinska University Hospital (Other); Tampere University (Other); Academy of Finland (Other); Uppsala University Hospital (Other); Aarhus University Hospital (Other); Regionaalhaigla, Tallinn (Unknown); Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Antti Launonen, MD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R10127
Record Dates: First submitted 2010-11-15; First posted 2010-11-23 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Humeral Fractures, Proximal
Keywords: Proximal humerus fracture; conservative; locking plate; Philos; Hemiprosthesis
MeSH Terms: conditions — Shoulder Fractures | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conservative (Active Comparator): Active physiotherapy and self-training
  Interventions: Other: Control group
- Philos locking plate (Active Comparator): After operative treatment active physiotherapy and self-training
  Interventions: Device: Philos
- Epoca prosthesis (Active Comparator): After operative treatment active physiotherapy and self-training
  Interventions: Device: Epoca

INTERVENTIONS:
Device: Philos — Conservative treatment versus Philos locking plate in 2 part fracture group.
  Conservative treatment versus Philos locking plating versus Epoca prosthesis in MFF group.
  Arms: Philos locking plate
Device: Epoca — Conservative treatment versus Philos locking plate versus Epoca fracture prosthesis in MFF group
  Arms: Epoca prosthesis
Other: Control group — Conservative control group
  Arms: Conservative

SUMMARY:
This trial is designed to compare head-to-head conservative with operative treatment in 2 stratum. Stratum 1: In 2 part fractures the comparison is between conservative treatment and operative treatment with plate fixation with Philos. Stratum 2: In multi-fragmented fractures (MFF) meaning 3 and 4 part fractures, the comparison is between conservative treatment, operative treatment with Philos plate and operative treatment with Epoca prosthesis. Subgroup analysis will be performed in an effort to obtain limit values for specific treatment of different age and fracture groups. A cost-effectiveness analysis and comparison between different treatment modalities will be carried out. The primary outcome measure will be the DASH score and the secondary outcome measure the EQ-5D value. Recruitment period is 3 years and follow-up 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Low energy proximal humeral displaced (more than 1 cm or 45 degrees) 2 part fracture where fracture line emerges through the surgical (or anatomical) neck
* Low energy proximal humeral displaced (more than 1 cm or 45 degrees) 3 or 4 part fracture

Exclusion Criteria:

* Refuse to participate the study
* Less than 60 years old
* Non-independent
* Dementia and/or institutionalized
* Does no understand written and spoken guidance in either Finnish or Swedish
* Pathological fracture or previous fracture in the same proximal humerus
* Serious intoxicant dependent, eg. In first aid breathalyzer shows more than 2‰
* Other operational injury in the same upper limb
* Major nerve injury (eg. Complete radialis- or delta palsy)
* Open fracture
* Multi-trauma or -fractured patient
* Fracture dislocation or head splitting fracture
* Undisplaced fracture
* Isolated tuberculum fracture
* Fracture has no precondition to ossify by conservative treatment (no bony contact between fracture parts or the humeral shaft is in contact with the articular surface)
* Treating surgeon considers patient unsuitable to attend the study on medical basis
* Cuff-arthropathy

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-01; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
DASH | 6 months
  to measure physical function and symptoms of the fractured shoulder
DASH | 1 year
  to measure physical function and symptoms of the fractured shoulder
DASH | 2 year
  to measure physical function and symptoms of the fractured shoulder

SECONDARY OUTCOMES:
EQ-5D | 6 month
  Individual's general health related quality of life is measured with EQ-5D
EQ-5D | 1 year
  Individual's general health related quality of life is measured with EQ-5D
EQ-5D | 2 year
  Individual's general health related quality of life is measured with EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Minna Laitinen, Docent, Principal Investigator — Tampere University Hospital; Antti Launonen, MD, Study Director — Tampere University Hospital; Pekka Rissanen, Professor, Study Chair — Tampere University; Johanna Ojanperä, MD, Study Chair — Kuopio University Hospital; Vesa Lepola, MD, PhD, Study Chair — Tampere University Hospital; Timo Viljakka, MD, Study Chair — Tampere University Hospital; Ville M Mattila, Professor, Study Chair — Tampere University Hospital; Juha Paloneva, MD PhD, Study Chair — Jyväskylä Central Hospital; Hans Berg, Docent, Study Chair — Karolinska University Hospital; Karl-Åke Jansson, Docent, Study Chair — Karolinska University Hospital; Kjeld Soballe, Professor, Study Chair — Aarhus University Hospital; Kaj Dossing, MD, Study Chair — Central Jutland Regional Hospital; Helle Ostergaard, Msc, Study Chair — Central Jutland Regional Hospital; Inger Mechlenburg, PhD, Study Chair — University of Aarhus
Locations (6):
- Aarhus University Hospital, Aarhus, Denmark
- Regionaalhaigla, PERH, Tallinn, Estonia
- Finland (2):
  - Jyväskylä Central Hospital, Jyväskylä, Central Finland
  - Tampere University Hospital, Tampere, Pirkanmaa
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Background] Launonen AP, Lepola V, Flinkkila T, Strandberg N, Ojanpera J, Rissanen P, Malmivaara A, Mattila VM, Elo P, Viljakka T, Laitinen M. Conservative treatment, plate fixation, or prosthesis for proximal humeral fracture. A prospective randomized study. BMC Musculoskelet Disord. 2012 Sep 7;13:167. doi: 10.1186/1471-2474-13-167. PMID 22954329
- [Derived] Launonen AP, Sumrein BO, Reito A, Lepola V, Paloneva J, Berg HE, Fellander-Tsai L, Kask K, Rahnel T, Tootsi K, Martson A, Jonsson KB, Wolf O, Strom P, Dossing K, Ostergaard HK, Mechlenburg I, Mattila VM, Laitinen MK. Surgery with locking plate or hemiarthroplasty versus nonoperative treatment of 3-4-part proximal humerus fractures in older patients (NITEP): An open-label randomized trial. PLoS Med. 2023 Nov 28;20(11):e1004308. doi: 10.1371/journal.pmed.1004308. eCollection 2023 Nov. PMID 38015877
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- [Derived] Launonen AP, Sumrein BO, Reito A, Lepola V, Paloneva J, Jonsson KB, Wolf O, Strom P, Berg HE, Fellander-Tsai L, Jansson KA, Fell D, Mechlenburg I, Dossing K, Ostergaard H, Martson A, Laitinen MK, Mattila VM; as the NITEP group. Operative versus non-operative treatment for 2-part proximal humerus fracture: A multicenter randomized controlled trial. PLoS Med. 2019 Jul 18;16(7):e1002855. doi: 10.1371/journal.pmed.1002855. eCollection 2019 Jul. PMID 31318863